CLINICAL TRIAL: NCT02446990
Title: Effects of Ivabradine in Patients With Stable Coronary Artery Disease Without Clinical Heart Failure. A Randomised Double-blind Placebo-controlled International Multicenter Study. Study Assessing the Morbi-mortality Benefits of the If Inhibitor Ivabradine in Patients With Coronary Artery Disease
Brief Title: Effects of Ivabradine in Patients With Stable Coronary Artery Disease Without Clinical Heart Failure
Acronym: SIGNIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-16257-083; 2009-011360-10 (EudraCT Number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-18 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Experimental)
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — 5 mg, 7.5 mg or 10 mg tablets to be taken orally twice daily, at 12-hours intervals, in the morning and in the evening during meals up to 48 months.
  Arms: Ivabradine
Drug: Placebo — Matching placebo tablets to be taken orally twice daily, at 12-hours intervals, in the morning and in the evening during meals up to 48 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of ivabradine on cardiovascular events in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of coronary artery disease
* Sinus rhythm and resting heart rate equal or higher than 70 bpm

Exclusion Criteria:

* Unstable cardiovascular condition
* Known hypersensitivity to ivabradine or current treatment with marketed ivabradine

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19102 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Italy
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Fox K, Ford I, Steg PG, Tardif JC, Tendera M, Ferrari R; SIGNIFY Investigators. Ivabradine in stable coronary artery disease without clinical heart failure. N Engl J Med. 2014 Sep 18;371(12):1091-9. doi: 10.1056/NEJMoa1406430. Epub 2014 Aug 31. PMID 25176136
- [Result] Fox K, Ford I, Steg PG, Tardif JC, Tendera M, Ferrari R. Rationale, design, and baseline characteristics of the Study assessInG the morbidity-mortality beNefits of the If inhibitor ivabradine in patients with coronarY artery disease (SIGNIFY trial): a randomized, double-blind, placebo-controlled trial of ivabradine in patients with stable coronary artery disease without clinical heart failure. Am Heart J. 2013 Oct;166(4):654-661.e6. doi: 10.1016/j.ahj.2013.06.024. Epub 2013 Sep 17. PMID 24093844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1181 centres in 51 countries screened at least one patient and 1139 centres included at least one patient.
Pre-assignment Details: A total of 23 164 patients were screened, 21 862 were selected and 19 107 were included. The Randomised Set comprised 19 102 patients: 9550 patients in the ivabradine group and 9552 in the placebo group. Of the 19 102 patients in the Randomised Set, 17 724 completed the study: 8830 patients in the ivabradine group and 8894 in the placebo group.
Period: Overall Study
Arm/Group | Ivabradine | Placebo
Started | 9550 | 9552
Completed | 8830 | 8894
Not Completed | 720 | 658
Not completed — Death | 485 | 458
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 231 | 199

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine | Placebo | Total
Number analyzed (Participants) | 9550 | 9552 | 19102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5109 | 5096 | 10205
  >=65 years | 4441 | 4456 | 8897
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.2) | 65 (7.3) | 65 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2601 | 2662 | 5263
  Male | 6949 | 6890 | 13839

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Endpoint
Description: First event among cardiovascular death or non-fatal myocardial infarction
Time Frame: The events are expressed as the time to occurrence of the first event, defined as the duration between the date of randomisation and the date of first occurrence of event, assessed up to 48 months.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 654 | 611
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.1969, Regression, Cox; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.96 to 1.2], Standard Error of Mean 0.06

2. Secondary Outcome: All-cause Mortality
Time Frame: From the date of randomisation to death, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 485 | 458
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.3461, Regression, Cox; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.94 to 1.21], Standard Error of Mean 0.07

3. Secondary Outcome: Cardiovascular Mortality
Description: Component of the primary composite endpoint
Time Frame: From the date of randomisation to death, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 329 | 301
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.2493, Regression, Cox; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.94 to 1.28], Standard Error of Mean 0.09

4. Secondary Outcome: Coronary Mortality
Description: Coronary mortality including sudden death of unknown cause, death from myocardial infarction, death from heart failure, death from coronary artery procedure, presumed arrhythmic death
Time Frame: From the date of randomisation to death, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 263 | 249
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.5162, Regression, Cox; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.89 to 1.26], Standard Error of Mean 0.09

5. Secondary Outcome: Fatal Myocardial Infarction
Description: Non-composite secondary endpoint
Time Frame: From the date of randomisation to death, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 51 | 38
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.1647, Regression, Cox; Cox Proportional Hazard = 1.35, 95% CI 2-sided [0.88 to 2.05], Standard Error of Mean 0.29

6. Secondary Outcome: Non-fatal Myocardial Infarction
Description: Component of the primary composite endpoint
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 351 | 339
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.6024, Regression, Cox; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.90 to 1.21], Standard Error of Mean 0.08

7. Secondary Outcome: Elective Coronary Revascularisation
Description: Non-composite secondary endpoint
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 270 | 305
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.1458, Regression, Cox; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.75 to 1.04]

8. Secondary Outcome: Coronary Revascularisation (Elective or Not)
Description: Non-composite secondary endpoint
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 562 | 564
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.9790, Regression, Cox; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.89 to 1.12]

9. Secondary Outcome: Secondary Composite Endpoint
Description: Fatal or non-fatal myocardial infarction
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 392 | 372
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.4299, Regression, Cox; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.92 to 1.22]

10. Secondary Outcome: Secondary Composite Endpoint
Description: Fatal or non-fatal myocardial infarction, coronary revascularisation
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 718 | 739
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.5916, Regression, Cox; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.88 to 1.08]

11. Secondary Outcome: Secondary Composite Endpoint
Description: Fatal or non-fatal myocardial infarction, coronary revascularisation, unstable angina
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 766 | 782
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.6963, Regression, Cox; Cox Proportional Hazard = 0.98, 95% CI 2-sided [0.89 to 1.08]

12. Secondary Outcome: Secondary Composite Endpoint
Description: Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 774 | 731
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.2222, Regression, Cox; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.96 to 1.18]

13. Secondary Outcome: Secondary Composite Endpoint
Description: Coronary death, non-fatal myocardial infarction
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 590 | 562
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.3671, Regression, Cox; Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.94 to 1.18]

14. Secondary Outcome: Secondary Composite Endpoint
Description: Non-fatal myocardial infarction, coronary revascularisation, unstable angina
Time Frame: From the date of randomisation to the date of first occurrence of the event, up to 48 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 9550 | 9552
participants | 734 | 759
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.5285, Regression, Cox; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.87 to 1.07]

ADVERSE EVENTS:
Time Frame: From randomisation to death, up to 48 months
Description: The Randomised Set consisted of 19 102 patients (9550 patients in the ivabradine group and 9552 in the placebo group). The Safety Set consisted of 19 083 patients: 19 randomised patients were excluded from the Safety Set because they did not take any study medication (11 patients in the ivabradine group and 8 in the placebo group).
Arm/Group | Ivabradine | Placebo
Serious Adverse Events (participants affected / at risk) | 3379/9539 | 3263/9544
Other Adverse Events (participants affected / at risk) | 6207/9539 | 5525/9544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=9539) | Placebo (N=9544)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 30 (30) | 45 (45)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 14 (14) | 15 (15)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 8 (8) | 0 (0)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 (7) | 8 (8)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Platelet dysfunction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (17) | 12 (12)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 17 (18) | 21 (24)
Acute left ventricular failure (Cardiac disorders) | 2 (3) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 200 (216) | 208 (229)
Adams-Stokes syndrome (Cardiac disorders) | 0 (0) | 3 (3)
Angina pectoris (Cardiac disorders) | 294 (314) | 330 (361)
Angina unstable (Cardiac disorders) | 409 (479) | 433 (524)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 3 (3) | 2 (2)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 12 (12) | 9 (9)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 336 (381) | 232 (262)
Atrial flutter (Cardiac disorders) | 49 (52) | 41 (45)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 17 (17) | 13 (13)
Atrioventricular block first degree (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 22 (22) | 13 (13)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 101 (102) | 21 (21)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 7 (7) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 5 (5) | 9 (9)
Cardiac arrest (Cardiac disorders) | 15 (16) | 8 (8)
Cardiac asthma (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure (Cardiac disorders) | 357 (415) | 346 (394)
Cardiac failure acute (Cardiac disorders) | 37 (45) | 23 (26)
Cardiac failure chronic (Cardiac disorders) | 25 (28) | 29 (36)
Cardiac failure congestive (Cardiac disorders) | 31 (33) | 24 (26)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 30 (30) | 22 (22)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 4 (4)
Cor pulmonale (Cardiac disorders) | 6 (6) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 20 (21) | 25 (25)
Coronary artery dissection (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 14 (14) | 7 (7)
Coronary artery stenosis (Cardiac disorders) | 18 (19) | 26 (26)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Endocarditis noninfective (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 5 (5) | 9 (9)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (5) | 6 (6)
Left atrial dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 3 (3)
Left ventricular failure (Cardiac disorders) | 9 (10) | 10 (10)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 16 (16) | 14 (14)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial depression (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 98 (104) | 83 (88)
Myocardial ischaemia (Cardiac disorders) | 23 (23) | 27 (27)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Nodal rhythm (Cardiac disorders) | 5 (5) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2) | 4 (4)
Pericardial effusion (Cardiac disorders) | 1 (1) | 5 (5)
Pericarditis (Cardiac disorders) | 3 (3) | 8 (8)
Postinfarction angina (Cardiac disorders) | 1 (1) | 2 (2)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 2 (2)
Rhythm idioventricular (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 8 (8) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 9 (9) | 5 (5)
Silent myocardial infarction (Cardiac disorders) | 5 (5) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 3 (3)
Sinus arrest (Cardiac disorders) | 9 (9) | 9 (9)
Sinus arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 48 (49) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 6 (6) | 12 (12)
Supraventricular extrasystoles (Cardiac disorders) | 8 (8) | 15 (15)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 17 (18) | 21 (24)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 6 (6) | 5 (5)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 32 (32) | 21 (21)
Ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 20 (20) | 20 (22)
Ventricular tachycardia (Cardiac disorders) | 35 (39) | 21 (23)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Metabolic myopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 9 (9) | 7 (9)
Vestibular ataxia (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 2 (2) | 3 (3)
Basedow's disease (Endocrine disorders) | 2 (2) | 2 (2)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Empty sella syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 4 (4) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 6 (7) | 5 (5)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 4 (4) | 4 (4)
Amaurosis (Eye disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 2 (2) | 4 (4)
Angle closure glaucoma (Eye disorders) | 1 (1) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 3 (3)
Blindness unilateral (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 39 (43) | 32 (32)
Cataract diabetic (Eye disorders) | 1 (1) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Choroidal effusion (Eye disorders) | 1 (1) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Dacryoadenitis acquired (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1)
Diabetic glaucoma (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 9 (9) | 18 (20)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 2 (3)
Glaucoma (Eye disorders) | 20 (20) | 19 (19)
Glaucomatous optic disc atrophy (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 1 (1)
Macular degeneration (Eye disorders) | 7 (8) | 6 (6)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 2 (2) | 1 (1)
Normal tension glaucoma (Eye disorders) | 2 (2) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 3 (3) | 4 (4)
Ophthalmoplegia (Eye disorders) | 0 (0) | 1 (1)
Optic atrophy (Eye disorders) | 0 (0) | 2 (2)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 28 (31) | 3 (3)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Retinal aneurysm (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 2 (2) | 4 (4)
Retinal artery thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 4 (4) | 6 (6)
Retinal haemorrhage (Eye disorders) | 10 (10) | 4 (4)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 3 (3)
Retinal vein thrombosis (Eye disorders) | 2 (2) | 0 (0)
Retinopathy haemorrhagic (Eye disorders) | 1 (1) | 1 (1)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 2 (2)
Retinoschisis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 13 (14) | 5 (5)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 3 (3)
Vitreous detachment (Eye disorders) | 3 (3) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 8 (10) | 4 (4)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 8 (8)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dental alveolar anomaly (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 9 (9)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 (4) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 7 (7) | 11 (11)
Duodenal ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 3 (3) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 8 (8) | 8 (8)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 10 (12) | 15 (16)
Gastric ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 14 (14) | 13 (13)
Gastritis atrophic (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastritis erosive (Gastrointestinal disorders) | 10 (10) | 10 (10)
Gastritis haemorrhagic (Gastrointestinal disorders) | 5 (5) | 7 (7)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (13) | 11 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (12) | 9 (10)
Gastrooesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 7 (7) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 (4) | 7 (7)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 7 (7) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 3 (3)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 29 (31) | 18 (18)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal angina (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 2 (2)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 11 (11) | 3 (3)
Leukoplakia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 3 (3)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 6 (6) | 4 (4)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mikulicz's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (12) | 8 (8)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral submucosal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 9 (9) | 17 (19)
Pancreatitis chronic (Gastrointestinal disorders) | 11 (11) | 7 (7)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Periproctitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 8 (8)
Rectal polyp (Gastrointestinal disorders) | 3 (3) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 3 (3) | 2 (2)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 6 (6)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8) | 7 (7)
Varices oesophageal (Gastrointestinal disorders) | 4 (4) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9) | 11 (11)
Apparent death (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 6 (6)
Cardiac death (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 3 (3) | 4 (4)
Chest pain (General disorders) | 32 (35) | 36 (50)
Chills (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 10 (10) | 7 (7)
Device breakage (General disorders) | 1 (1) | 1 (1)
Device dislocation (General disorders) | 3 (3) | 2 (2)
Device extrusion (General disorders) | 1 (1) | 0 (0)
Device failure (General disorders) | 2 (2) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Drug interaction (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 4 (4)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Foreign body reaction (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 3 (3) | 2 (2)
Generalised oedema (General disorders) | 3 (5) | 2 (2)
Hernia obstructive (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 3 (3)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 5 (5) | 8 (8)
Non-cardiac chest pain (General disorders) | 38 (43) | 29 (31)
Oedema peripheral (General disorders) | 9 (9) | 6 (6)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Spinal pain (General disorders) | 3 (4) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 43 (43) | 46 (46)
Sudden death (General disorders) | 75 (75) | 74 (74)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 4 (4) | 4 (4)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 3 (3)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 6 (6)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 9 (10) | 10 (10)
Cholecystitis acute (Hepatobiliary disorders) | 19 (19) | 17 (17)
Cholecystitis chronic (Hepatobiliary disorders) | 7 (7) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 12 (12) | 20 (20)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Chronic hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 7 (8) | 4 (4)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 4 (4)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 3 (3) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 2 (2)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 16 (18) | 9 (9)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 3 (3)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 2 (2) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 16 (16) | 22 (28)
Bronchitis bacterial (Infections and infestations) | 4 (4) | 0 (0)
Bronchopneumonia (Infections and infestations) | 29 (33) | 24 (26)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Candida pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 23 (23) | 18 (19)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholangitis suppurative (Infections and infestations) | 0 (0) | 2 (2)
Cholecystitis infective (Infections and infestations) | 5 (5) | 3 (3)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 4 (4) | 4 (5)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 4 (4)
Diabetic foot infection (Infections and infestations) | 5 (6) | 8 (8)
Diabetic gangrene (Infections and infestations) | 4 (4) | 13 (15)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 5 (5) | 8 (9)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Echinococciasis (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis enterococcal (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Epiglottitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 20 (20) | 15 (15)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 7 (7)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 7 (9) | 5 (5)
Gastroenteritis (Infections and infestations) | 16 (16) | 16 (16)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (3)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 2 (2) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 3 (3)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster ophthalmic (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 3 (4)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 3 (4) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 (5) | 6 (7)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Keratitis herpetic (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Legionella infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 3 (3) | 1 (1)
Lobar pneumonia (Infections and infestations) | 6 (6) | 13 (13)
Localised infection (Infections and infestations) | 0 (0) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 9 (10)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 4 (4) | 1 (1)
Lung infection (Infections and infestations) | 11 (11) | 8 (11)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Orchitis (Infections and infestations) | 2 (2) | 3 (3)
Osteomyelitis (Infections and infestations) | 2 (2) | 11 (11)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 2 (4)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perihepatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 9 (9) | 9 (9)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 122 (129) | 102 (112)
Pneumonia bacterial (Infections and infestations) | 7 (8) | 7 (7)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 2 (2)
Postoperative abscess (Infections and infestations) | 0 (0) | 3 (3)
Postoperative wound infection (Infections and infestations) | 6 (6) | 12 (13)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculoma (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 4 (4) | 1 (1)
Puncture site abscess (Infections and infestations) | 0 (0) | 1 (1)
Puncture site infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 5 (5) | 8 (8)
Pyelonephritis chronic (Infections and infestations) | 7 (7) | 6 (8)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Renal tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 5 (5) | 12 (13)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 11 (11) | 11 (11)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 9 (9) | 13 (13)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Small intestine gangrene (Infections and infestations) | 0 (0) | 1 (1)
Sputum purulent (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 4 (4) | 2 (2)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 3 (3) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 1 (1) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 2 (2) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 26 (26) | 17 (18)
Urinary tract infection bacterial (Infections and infestations) | 7 (7) | 3 (3)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 13 (14)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection bacterial (Infections and infestations) | 3 (3) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Agitation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asbestosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blindness traumatic (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Concussion (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 9 (9) | 8 (8)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 9 (9) | 12 (12)
Corrosive gastritis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
Crushing injury of trunk (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 95 (96) | 109 (109)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 13 (13) | 12 (12)
Femur fracture (Injury, poisoning and procedural complications) | 15 (15) | 10 (10)
Fibula fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 10 (11)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 14 (14) | 13 (14)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-thoracotomy pain syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 8 (8) | 15 (15)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 8 (8) | 15 (15)
Road traffic accident (Injury, poisoning and procedural complications) | 23 (23) | 26 (26)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Silicosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Skull fractured base (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 8 (8) | 7 (7)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Suture related complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 11 (11) | 11 (11)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Arteriogram carotid (Investigations) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 43 (45) | 53 (58)
Arthroscopy (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 12 (12) | 10 (10)
Biopsy prostate (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 6 (6)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood parathyroid hormone decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 4 (4) | 1 (1)
Blood pressure decreased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 24 (26) | 13 (14)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Carbohydrate antigen 19-9 increased (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Cardiovascular evaluation (Investigations) | 78 (98) | 84 (100)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1) | 0 (0)
Cystoscopy normal (Investigations) | 0 (0) | 1 (1)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 57 (60) | 18 (18)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ambulatory (Investigations) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Gastrointestinal examination (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 6 (6)
Heart rate decreased (Investigations) | 55 (55) | 7 (7)
Hepatic enzyme increased (Investigations) | 2 (2) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 3 (3)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1)
Investigation (Investigations) | 7 (7) | 6 (7)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Pulmonary arterial pressure increased (Investigations) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0)
Romberg test positive (Investigations) | 0 (0) | 1 (1)
Sleep study (Investigations) | 3 (3) | 1 (1)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0)
Stress echocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1) | 0 (0)
Treponema test positive (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 11 (11)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 19 (20) | 19 (19)
Diabetes mellitus (Metabolism and nutrition disorders) | 59 (65) | 82 (87)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 34 (36) | 50 (53)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (11) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (14) | 10 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 19 (20) | 12 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 25 (26) | 47 (52)
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 (12) | 20 (20)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 46 (47) | 43 (48)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (10)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 (18) | 16 (18)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 7 (7)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (25) | 21 (23)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 9 (9)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Bladder cancer stage I, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Chronic lymphocytic leukaemia stage 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Clear cell sarcoma of soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 8 (8)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Large cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lip and/or oral cavity cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (9)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 10 (10)
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 12 (12)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of choroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 8 (8)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Penis carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pineal parenchymal neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 (38) | 18 (18)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Urethral cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 5 (5) | 2 (2)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 2 (2)
Anticholinergic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 4 (4)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid aneurysm rupture (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 4 (4) | 3 (3)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery disease (Nervous system disorders) | 2 (2) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 3 (3) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 51 (57) | 43 (45)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 4 (4)
Carpal tunnel syndrome (Nervous system disorders) | 4 (4) | 6 (6)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 4 (4) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral infarction (Nervous system disorders) | 15 (15) | 13 (13)
Cerebral ischaemia (Nervous system disorders) | 8 (9) | 3 (3)
Cerebral microangiopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 31 (32) | 40 (44)
Cerebrovascular disorder (Nervous system disorders) | 5 (5) | 3 (3)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 2 (2)
Coma (Nervous system disorders) | 2 (2) | 3 (3)
Convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 4 (4) | 4 (4)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Dementia of the Alzheimer's type, with delusions (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 10 (10) | 10 (10)
Dizziness (Nervous system disorders) | 19 (19) | 18 (20)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2) | 2 (2)
Dystonic tremor (Nervous system disorders) | 1 (1) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Encephalomyelitis (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 4 (4) | 2 (2)
Epilepsy (Nervous system disorders) | 7 (9) | 5 (5)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 4 (4) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 5 (6) | 12 (12)
Headache (Nervous system disorders) | 5 (5) | 8 (8)
Hemianopia homonymous (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 6 (7) | 1 (1)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 2 (2) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 9 (10)
Hypoglycaemic coma (Nervous system disorders) | 2 (3) | 5 (5)
Hypoglycaemic unconsciousness (Nervous system disorders) | 4 (4) | 9 (9)
Hyporeflexia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 4 (4) | 5 (5)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 97 (100) | 90 (95)
Lacunar infarction (Nervous system disorders) | 5 (5) | 6 (6)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 32 (32) | 22 (22)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 4 (4)
Memory impairment (Nervous system disorders) | 4 (4) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root lesion (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 1 (1)
Neuritis cranial (Nervous system disorders) | 0 (0) | 2 (2)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (2)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 6 (6) | 8 (8)
Parkinsonism (Nervous system disorders) | 2 (2) | 3 (3)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 4 (4)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1)
Post-injection delirium sedation syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 15 (15) | 8 (8)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Radial nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 2 (2)
Radicular syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Radiculopathy (Nervous system disorders) | 5 (5) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Retrograde amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 8 (9)
Senile dementia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 1 (1)
Spinal vascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 3 (3)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 91 (102) | 89 (96)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Tonic convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 56 (59) | 50 (50)
Tremor (Nervous system disorders) | 0 (0) | 3 (3)
Ulnar neurapraxia (Nervous system disorders) | 0 (0) | 1 (1)
Ulnar tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 2 (2)
VIth nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Vascular dementia (Nervous system disorders) | 3 (3) | 3 (3)
Vascular encephalopathy (Nervous system disorders) | 11 (11) | 9 (9)
Vertebral artery occlusion (Nervous system disorders) | 2 (2) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 3 (3) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 15 (15) | 12 (16)
Vertigo CNS origin (Nervous system disorders) | 2 (2) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0)
Wernicke-Korsakoff syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 3 (3) | 2 (2)
Agitated depression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 4 (4)
Confusional state (Psychiatric disorders) | 7 (7) | 10 (10)
Delirium (Psychiatric disorders) | 8 (9) | 7 (7)
Delirium tremens (Psychiatric disorders) | 1 (1) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 57 (59) | 54 (54)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 3 (3)
Dysthymic disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Intentional drug misuse (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 1 (2)
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Obsessive thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Persecutory delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosomatic disease (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 3 (4)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Anuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck sclerosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (2)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 7 (7) | 6 (6)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 10 (10) | 7 (7)
Cystitis glandularis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 4 (4) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 11 (12) | 7 (7)
Dysuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 6 (6) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 5 (6)
Hydroureter (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephroangiosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 7 (7) | 14 (14)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 6 (6) | 3 (3)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 38 (39) | 30 (30)
Renal failure acute (Renal and urinary disorders) | 29 (31) | 35 (38)
Renal failure chronic (Renal and urinary disorders) | 34 (35) | 17 (17)
Renal impairment (Renal and urinary disorders) | 13 (14) | 5 (5)
Renal infarct (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal ischaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 3 (3) | 6 (6)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 12 (14) | 18 (18)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Acquired phimosis (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 23 (23) | 28 (28)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 31 (33) | 30 (32)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 12 (13)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 16 (21)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (5)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 64 (84) | 52 (62)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 23 (26)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 24 (24)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (5)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 10 (10)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 12 (12)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 27 (28)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (10)
Dry gangrene (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (11)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Activities of daily living impaired (Social circumstances) | 11 (11) | 1 (1)
Alcohol use (Social circumstances) | 2 (2) | 0 (0)
Immobile (Social circumstances) | 1 (1) | 0 (0)
Impaired driving ability (Social circumstances) | 15 (15) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Aortic valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 3 (3)
Arterial bypass operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardiac aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 23 (30) | 19 (27)
Carotid angioplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Carotid artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid artery stent insertion (Surgical and medical procedures) | 2 (2) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 2 (2) | 3 (3)
Cataract operation (Surgical and medical procedures) | 9 (9) | 9 (10)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 1 (2)
Cholecystectomy (Surgical and medical procedures) | 6 (6) | 2 (2)
Cholesteatoma removal (Surgical and medical procedures) | 1 (2) | 0 (0)
Circumcision (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 5 (5)
Coronary arterial stent insertion (Surgical and medical procedures) | 5 (5) | 2 (2)
Coronary artery bypass (Surgical and medical procedures) | 10 (10) | 18 (18)
Coronary revascularisation (Surgical and medical procedures) | 8 (8) | 5 (5)
Diabetes mellitus management (Surgical and medical procedures) | 4 (5) | 8 (12)
Dupuytren's contracture operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Fasciectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Femoral hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Finger amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric banding (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 2 (2)
Glaucoma surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 9 (10) | 9 (9)
Hospitalisation (Surgical and medical procedures) | 8 (13) | 10 (11)
Hydrocele operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ileostomy closure (Surgical and medical procedures) | 0 (0) | 2 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 2 (2) | 0 (0)
Incisional hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Infusion (Surgical and medical procedures) | 0 (0) | 3 (7)
Inguinal hernia repair (Surgical and medical procedures) | 3 (3) | 9 (9)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Keratoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 4 (4) | 12 (13)
Knee operation (Surgical and medical procedures) | 1 (1) | 2 (2)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Lens extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Liver operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 2 (2) | 1 (1)
Meniscus removal (Surgical and medical procedures) | 2 (2) | 0 (0)
Metatarsal excision (Surgical and medical procedures) | 0 (0) | 1 (2)
Mitral valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Obesity surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 15 (15) | 16 (16)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 4 (4)
Peripheral artery bypass (Surgical and medical procedures) | 2 (2) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Physiotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Radical hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 8 (12) | 10 (14)
Removal of internal fixation (Surgical and medical procedures) | 4 (4) | 1 (1)
Renal artery ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal stone removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Retinal laser coagulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 2 (2) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Suture insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 3 (3) | 2 (2)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 2 (2)
Urethral dilation procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary calculus removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Uterine polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginal prolapse repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 4 (4) | 7 (7)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 5 (5) | 2 (2)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 2 (2) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 7 (8) | 2 (2)
Circulatory collapse (Vascular disorders) | 2 (2) | 7 (8)
Deep vein thrombosis (Vascular disorders) | 19 (19) | 17 (17)
Diabetic macroangiopathy (Vascular disorders) | 1 (1) | 1 (1)
Diabetic microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 2 (2)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 5 (6) | 7 (7)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 10 (11) | 14 (15)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 204 (220) | 144 (152)
Hypertensive crisis (Vascular disorders) | 104 (117) | 105 (119)
Hypertensive emergency (Vascular disorders) | 13 (15) | 8 (8)
Hypotension (Vascular disorders) | 25 (26) | 36 (37)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 4 (4)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 4 (4)
Iliac artery rupture (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 5 (5) | 8 (9)
Jugular vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Labile blood pressure (Vascular disorders) | 1 (1) | 1 (1)
Labile hypertension (Vascular disorders) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Lymphostasis (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 12 (12) | 6 (6)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 52 (58) | 67 (70)
Peripheral artery aneurysm (Vascular disorders) | 3 (3) | 3 (3)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 13 (16) | 12 (12)
Peripheral artery thrombosis (Vascular disorders) | 6 (6) | 6 (6)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 8 (8)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 5 (5)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 3 (3) | 5 (6)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 5 (5) | 6 (6)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose ulceration (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 3 (3) | 2 (2)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Withdrawal hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=9539) | Placebo (N=9544)
Anaemia (Blood and lymphatic system disorders) | 186 (191) | 197 (204)
Angina pectoris (Cardiac disorders) | 340 (370) | 388 (413)
Atrial fibrillation (Cardiac disorders) | 135 (157) | 101 (108)
Atrioventricular block first degree (Cardiac disorders) | 247 (265) | 203 (221)
Bradycardia (Cardiac disorders) | 473 (511) | 57 (63)
Cardiac failure (Cardiac disorders) | 125 (131) | 132 (137)
Sinus bradycardia (Cardiac disorders) | 144 (150) | 15 (17)
Sinus tachycardia (Cardiac disorders) | 40 (40) | 161 (181)
Supraventricular extrasystoles (Cardiac disorders) | 176 (186) | 128 (129)
Ventricular extrasystoles (Cardiac disorders) | 310 (331) | 244 (267)
Cataract (Eye disorders) | 118 (132) | 158 (171)
Photopsia (Eye disorders) | 483 (536) | 48 (49)
Vision blurred (Eye disorders) | 102 (105) | 31 (31)
Constipation (Gastrointestinal disorders) | 95 (102) | 98 (102)
Diarrhoea (Gastrointestinal disorders) | 117 (121) | 112 (120)
Gastritis (Gastrointestinal disorders) | 96 (97) | 111 (114)
Chest pain (General disorders) | 79 (86) | 98 (108)
Fatigue (General disorders) | 119 (124) | 106 (112)
Oedema peripheral (General disorders) | 205 (225) | 165 (172)
Bronchitis (Infections and infestations) | 214 (241) | 182 (198)
Influenza (Infections and infestations) | 113 (123) | 168 (176)
Nasopharyngitis (Infections and infestations) | 172 (195) | 172 (198)
Upper respiratory tract infection (Infections and infestations) | 166 (194) | 175 (215)
Urinary tract infection (Infections and infestations) | 105 (111) | 100 (118)
Fall (Injury, poisoning and procedural complications) | 174 (188) | 194 (204)
Blood creatinine increased (Investigations) | 111 (115) | 88 (89)
Blood pressure increased (Investigations) | 95 (119) | 106 (131)
C-reactive protein increased (Investigations) | 154 (158) | 139 (142)
Electrocardiogram QT prolonged (Investigations) | 106 (118) | 40 (44)
Heart rate decreased (Investigations) | 985 (1118) | 105 (116)
Diabetes mellitus (Metabolism and nutrition disorders) | 185 (199) | 247 (260)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 155 (162) | 174 (183)
Hyperglycaemia (Metabolism and nutrition disorders) | 99 (102) | 99 (104)
Hyperkalaemia (Metabolism and nutrition disorders) | 140 (145) | 111 (121)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 150 (154) | 158 (161)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 136 (141) | 173 (179)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (74) | 96 (99)
Back pain (Musculoskeletal and connective tissue disorders) | 95 (100) | 108 (114)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 105 (116) | 155 (161)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 107 (113) | 118 (125)
Dizziness (Nervous system disorders) | 275 (292) | 202 (215)
Headache (Nervous system disorders) | 165 (190) | 139 (154)
Insomnia (Psychiatric disorders) | 98 (100) | 98 (101)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 98 (98) | 104 (104)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 113 (127) | 112 (136)
Cough (Respiratory, thoracic and mediastinal disorders) | 147 (158) | 137 (144)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 114 (119) | 93 (95)
Hypertension (Vascular disorders) | 968 (1102) | 810 (918)
Hypotension (Vascular disorders) | 155 (161) | 155 (161)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publication and/or communication related to the study results and can require changes. In case of a patent application, the sponsor can delay its authorization for publication or communication of the study results until the date of international registration of the patent.